CLINICAL TRIAL: NCT00216268
Title: Treatment of Japanese Encephalitis - a Double Blind Placebo Controlled Trial
Brief Title: Treatment of Japanese Encephalitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indian Council of Medical Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5/8/7/1/13/2001-ECD1
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2006-02-09 (Estimated); Status verified 2005-09

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Ribavirin

INTERVENTIONS:
Drug: Ribavirin

SUMMARY:
Japanese encephalitis is the single largest cause of viral encephalitis in the world today. It occurs in yearly post monsoon outbreaks in Uttar Pradesh and other parts of India and south east Asia. There is presently no antiviral drug of proven benefit for this illness and treatment is mostly supportive. The drug Ribavirin is already in the market in use for other indications. It has been found useful in West Nile encephalitis and various hemorrhagic fevers caused by related arboviruses. This is a double blind placebo of Ribavirin in Japanese encephalitis. To the best of our knowledge, this is the first such trial in the world. The study hypothesis is that children treated with ribavirin will be no different from those getting placebo in terms of mortality, length of hospital stay, days to return to consciousness and oral feeds, days to become afebrile and convulsion free and in 3 month sequelae rate.

ELIGIBILITY:
Inclusion Criteria:

* Child between 6 months and 12 years age
* Acute febrile encephalopathy
* Positive IgM ELISA test for Japanese encephalitis in serum

Exclusion Criteria:

* Consent not obtained

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Start 2005-07; Study Completion 2008-05

PRIMARY OUTCOMES:
Mortality during hospital stay

SECONDARY OUTCOMES:
Sequelae at 3 months
Duration of hospital stay
Days to return to oral feeds
Days to become convulsion free
Days to become afebrile

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Kumar, Principal Investigator — King George Medical University, Lucknow INDIA
Locations (1):
- King George Medical University, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Derived] Kumar R, Tripathi P, Baranwal M, Singh S, Tripathi S, Banerjee G. Randomized, controlled trial of oral ribavirin for Japanese encephalitis in children in Uttar Pradesh, India. Clin Infect Dis. 2009 Feb 15;48(4):400-6. doi: 10.1086/596309. PMID 19143532